CLINICAL TRIAL: NCT02119351
Title: A Post-market, Randomized Study Evaluating the Clinical Performance of the ViaValve™ Safety IV Catheter
Brief Title: A Study Evaluating the Clinical Performance of the ViaValve™ Safety IV Catheter
Acronym: ViaValve-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smiths Medical, ASD, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ViaValve Study
Record Dates: First submitted 2013-07-12; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Peripheral Intravenous Catheter
Keywords: peripheral intravenous catheters; blood exposure; blood control; IV catheter insertion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ViaValve™ Safety IV Catheter (Active Comparator): Insertion of the ViaValve™ Safety IV Catheter
  Interventions: Device: ViaValve™ Safety IV Catheter
- ProtectIV® Plus Safety IV Catheter (Active Comparator): Insertion of the ProtectIV® Plus Safety IV Catheter
  Interventions: Device: ProtectIV® Plus Safety IV Catheter

INTERVENTIONS:
Device: ViaValve™ Safety IV Catheter — Safety peripheral IV catheter with a blood control feature
  Arms: ViaValve™ Safety IV Catheter
Device: ProtectIV® Plus Safety IV Catheter — Safety peripheral IV catheter with no blood control feature
  Arms: ProtectIV® Plus Safety IV Catheter

SUMMARY:
The objective of this post-market, prospective study is to evaluate the clinical acceptability, blood leakage, risk for blood exposure, need for digital compression, insertion success, and clinical utility of the ViaValve™ Safety IV Catheter compared to standard hospital PIVCs currently being used.

ELIGIBILITY:
Inclusion Criteria:

* A peripheral intravenous catheter will need to be inserted in order to gain access to a vein or artery to sample blood, monitor blood pressure, or administer fluids intravenous infusion as part of treatment.
* Willing and able to sign an Informed Consent (patient or legally authorized representative).

Exclusion Criteria:

* Body morphology (e.g., size) precludes the use of a peripheral intravenous catheter.
* Fluid to be infused is not appropriate for peripheral intravenous catheters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical acceptability of PIVC insertion | Clinicians will provide the rating immediately after performing the insertion
  Demonstrate non-inferiority of the ViaValve™ Safety I.V. Catheter compared to the control PIVC for ratings of clinical acceptability. Clinicians will agree or disagree that the device was clinically acceptable for the insertion.
Frequency of blood leakage | Clinicians will report if blood leakage occurred immediately after the catheter insertion
  Demonstrate superiority of the ViaValve™ Safety I.V. Catheter compared to the control in preventing blood leakage from the catheter hub during insertion.
Eliminating risk of blood exposure | Clinicians will report on the ability of the PIVC to eliminate blood exposure immediately after catheter insertion
  Demonstrate superiority of the ViaValve™ Safety I.V. Catheter compared to the control PIVC in eliminating the clinician's risk of blood exposure during the insertion process.

SECONDARY OUTCOMES:
Insertion success | Clinicians will report if the insertion was successful immediately after performing insertion
  Demonstrate the insertion success rate of the ViaValve™ I.V. Catheter is non-inferior to the control PIVC. Insertion success defined as a catheter confirmed successfully placed within the selected vessel in 3 or fewer venipuncture attempts.
Elimination of digital compression | Clinicians will provide the rating immediately after performing the insertion
  Demonstrate that the ViaValve™ Safety I.V. Catheter is non-inferior to the control PIVC in eliminating the clinician's need to use digital compression during the insertion process. Clinicians will agree or disagree the device eliminates the need for digital compression after each PIVC insertion.
Ease of Use | Clinicians will provide the rating immediately after performing the insertion
  Demonstrate that the ViaValve™ Safety I.V. Catheter is non-inferior to the control PIVC in seven measures of ease of use. Clinicians will agree or disagree with seven statements regarding ease of use/clinical utility.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McRae, MD, PhD, Principal Investigator — U of Calgary and Alberta Health Services
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada